CLINICAL TRIAL: NCT04019197
Title: Effects of GLP-l Receptor Agonists on Cardiometabolic Alterations in HIV-associated Lipohypertrophy
Brief Title: Effects of Semaglutide in HIV-Associated Lipohypertrophy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Medical University of South Carolina (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Allison Eckard, Multiple Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20190121; R01DK121619 (NIH)
Record Dates: First submitted 2019-07-01; First posted 2019-07-15 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS; Lipohypertrophy; Obesity
Keywords: HIV; lipohypertrophy; semaglutide; GLP-1 receptor agonist; obesity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with HIV and lipohypertrophy: semaglutide arm (Experimental): Participants with HIV/lipohypertrophy will receive semaglutide 0.25 mg x4 weeks, then semaglutide 0.5 mg x4 weeks, then semaglutide 1.0 mg x24 weeks, then no drug x24 weeks.
  Interventions: Drug: Semaglutide Injectable Product
- Participants with HIV and lipohypertrophy: placebo arm (Placebo Comparator): Participants with HIV/Lipohypertrophy will receive placebo x32 weeks, then no placebo for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Injectable Product — semaglutide subcutaneous injection
  Other Names: semaglutide; Ozempic
  Arms: Participants with HIV and lipohypertrophy: semaglutide arm
Drug: Placebo — placebo injection
  Other Names: placebo injection; placebos
  Arms: Participants with HIV and lipohypertrophy: placebo arm

SUMMARY:
This is a randomized, double-blinded, placebo-controlled trial designed to assess the effect of the GLP-1 receptor agonist, semaglutide, on visceral and ectopic fat, insulin resistance, inflammation markers, and the downstream effect of cardiovascular risk in people with HIV. The primary endpoints will be visceral and ectopic fat changes over the study period. The secondary endpoints will include changes in markers of inflammation, immune activation, gut integrity, and cardiovascular disease risk assessment.

DETAILED DESCRIPTION:
This study is a phase IIb, randomized, double-blinded, placebo-controlled clinical trial of semaglutide in people with HIV-associated lipohypertrophy. Participants will be recruited from 1 site (Cleveland, OH). The duration of the study will be 56 weeks. The interventional phase will last 32 weeks, followed by a 24-week observational phase to assess the sustainability of the intervention. Participants will be randomized 1:1 to receive semaglutide by subcutaneous injection once weekly for 32 weeks (8-week dose escalation phase followed by full-dose for 24 weeks) or matching placebo. The primary objective of this clinical trial is to determine the efficacy of semaglutide in treating lipohypertrophy among non-diabetic people living with HIV by reducing fat accumulation and ectopic fat deposition, altering adipokine levels, improving endothelial function and arterial stiffness, down-regulating key pro-inflammatory cytokines and immune activation without modifying microbial translocation and gut integrity markers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years.
2. HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
3. Body mass index ≥25 kg/m2.
4. Waist circumference and waist-to-hip ratio >95 cm and >0.94 cm, respectively, for men, and >94 cm and >0.88 cm, respectively, for women occurring in the context of HIV treatment.
5. Subjective evidence of increased abdominal girth occurring after initiation of HIV treatment.
6. HIV-1 RNA <400 copies/mL for ≥6 months.
7. Receiving a stable antiretroviral regimen for at least the last 12 weeks prior to study entry with cumulative duration of 1 year of treatment at the time of study entry.
8. Provision of signed and dated informed consent form and is capable of reading and comprehending the informed consent.
9. Stated willingness to comply with all study procedures and availability for the duration of the study.
10. All women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to start of study medication. WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), who is not postmenopausal (defined as amenorrhea 12 consecutive months), or is on hormone replacement therapy (HRT) with documented plasma follicle-stimulating hormone level 35 mIU/mL. Women who are using oral, implanted, or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), should be considered of child-bearing potential.
11. Female subjects who are not of reproductive potential (have reached menopause or undergone hysterectomy, bilateral oophorectomy or tubal ligation) or whose male partner has undergone successful vasectomy with resulting azoospermia or has azoospermia for any other reason, are eligible without requiring the use of contraception. Patient-reported history of menopause, sterilization, and azoospermia is considered acceptable documentation.
12. All subjects must not participate in a conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female subject/male partner must use condoms (male or female) in addition to one of the following forms of contraception while on study: either a spermicidal agent, diaphragm, cervical cap, IUD, or hormonal-based contraception.
13. Have no plans to alter antiretroviral therapy, or to undergo any weight loss program, formal exercise training or surgery during the study period, or initiate structured/strategic antiretroviral treatment interruptions.

Exclusion Criteria:

1. Known cardiovascular disease or diagnosed diabetes. If on metformin without a diabetes diagnoses metformin use has to be constant, uninterrupted for 6 months prior to entry.
2. Any active or chronic uncontrolled inflammatory condition, infection or cancer.
3. Women who are pregnant or breastfeeding.
4. Women with a positive pregnancy test on enrollment or prior to study drug administration.
5. A clinically-relevant illness within 14 days prior to study entry not explicitly excluded by the protocol, a physical or psychiatric disability, or a laboratory abnormality that might place the subject at increased risk by being exposed to the medications in this study or which might confound the interpretation of this investigation.
6. Active gastrointestinal symptom Grade >1 within the last month.
7. Regular use of immunomodulators/agents which could impact inflammation. Regular use of NSAIDS allowed if constant, uninterrupted for 6 months and no plans to alter. Statin use must also be constant, uninterrupted for 6 months prior to study entry. Thyroid medication allowed unless diagnosed with uncontrolled thyroid disease.
8. Inability to communicate effectively with study personnel.
9. Use of megestrol acetate, testosterone, or any steroid use beyond normal amounts found in the body within 6 months of study, or intend to start.
10. Glomerular filtration rate <50 cc/min/1.73 m2.
11. Hemoglobin <10 g/dL.
12. Elevated lipase level >1.5 upper limit of normal
13. AST AND ALT >2.5x upper limit of normal.
14. Use of growth hormone or growth hormone-releasing hormone in the last year, or intent to start.
15. History of excessive alcohol use (on average 2 or more drinks a day) , pancreatitis, thyroid cancer, or a diagnosis of multiple endocrine neoplasia (MEN) syndrome type 2.
16. History of lactose intolerance or inability to consume milk products will be exclusionary for participation in the mixed-meal tolerance test portion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Effects of semaglutide on quantity of abdominal fat (total, subcutaneous, visceral) | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the amount of abdominal fat (total, subcutaneous, visceral) as measured in area via abdominal CT scan.
Effects of semaglutide on quantity of fat (total body fat, limb fat, trunk fat) | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the amount of abdominal fat (total, subcutaneous, visceral) as measured in mass via whole-body DXA scan.
Effects of semaglutide on quantity of pericardial fat | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the amount of pericardial fat as measured in volume by chest CT scan.

SECONDARY OUTCOMES:
Effects of semaglutide on liver fat | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on liver fat as measured by density via abdominal CT scan.
Effects of semaglutide on quantity of lean body mass | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the amount of lean body mass as measured by whole-body DXA scan.
Effects of semaglutide on quantity of total right psoas muscle | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the amount of total right psoas muscle as measured in area via CT scan.
Effects of semaglutide on quality of abdominal fat (total, subcutaneous, visceral) | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the quality of abdominal fat (total, subcutaneous, visceral) as measured by density via CT scan.
Effects of semaglutide on quality of pericardial fat | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the quality of pericardial fat (total, subcutaneous, visceral) as measured by density via abdominal CT scan.
Effects of semaglutide on quality of total right psoas muscle | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on the quality/intermuscular fat content of total right psoas muscle as measured by density via CT scan.
Effects of semaglutide on anthropometric measurements (weight, waist circumference, waist-to-hip ratio) | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on anthropometric measurements.
Effects of semaglutide on glucose metabolism | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on on glucose metabolism by assessing oral glucose tolerance, fasting glucose levels, and HgbA1C.
Effects of semaglutide on lipoprotein profiles | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on lipoprotein profiles and oxidized LDL levels.
Effects of semaglutide on systemic inflammation | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on soluble markers of inflammation and immune activation to assess overall level of systemic inflammation.
Effects of semaglutide on systemic immune activation | 32 weeks
  Effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on cellular markers of inflammation and immune activation markers to assess overall level of systemic immune activation.
Effects of semaglutide on insulin sensitivity/resistance | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on insulin sensitivity/insulin resistance by assessing insulin levels, HOMA-IR (calculated based on insulin levels and glucose levels), and timed insulin levels as part of a 4-hour mixed meal tolerance test.
Effects of semaglutide on gut hormones | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in the gut hormones, GIP and GLP-1 levels, by means of a 4-hour mixed-meal tolerance test.
Effects of semaglutide on gut integrity | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in select measures of gut integrity and microbial translocation (e.g., I-FABP, zonulin-1, LPS).
Effects of semaglutide on resting energy expenditure | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in resting energy expenditure by means of indirect calorimetry.
Effects of semaglutide on pulse wave velocity | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in pulse wave velocity, a measure of arterial stiffness, as a surrogate measure of cardiovascular disease risk.
Effects of semaglutide on EndoPat | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in EndoPat, a measure of endothelial function, as a surrogate measure of cardiovascular disease risk.
Effects of semaglutide on coronary artery calcium (CAC) score | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in coronary artery calcium (CAC) score as measured by chest CT scan.
Effects of semaglutide on overall cardiovascular disease (CVD) risk | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, in overall cardiovascular disease (CVD) risk.
Effects of semaglutide on bone | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on bone markers and total bone mineral content as measured by whole-body DXA scan.
Effects of semaglutide on dietary intake | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on dietary intake via comprehensive dietary intake assessments.
Effects of semaglutide on physical activity | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on physical activity status via comprehensive physical activity assessments.
Safety analyses | 32 weeks
  Safety of semaglutide in HIV will be investigated, including a comparison between participants receiving semaglutide vs. placebo, on adverse events, side effects, and related safety endpoints.
Sustainability of effects of semaglutide on quantity of abdominal fat (total, subcutaneous, visceral) | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the amount of abdominal fat (total, subcutaneous, visceral) as measured in area via abdominal CT scan.
Sustainability of effects of semaglutide on quantity of fat (total body fat, limb fat, trunk fat) | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the amount of total fat, limb fat, and trunk fat as measured in mass via whole-body DXA scan.
Sustainability of effects of semaglutide on quantity of pericardial fat | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the amount of pericardial fat as measured in volume by chest CT scan.
Sustainability of effects of semaglutide on liver fat | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on liver fat as measured by density via abdominal CT scan.
Sustainability of effects of semaglutide on quantity of lean body mass | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the amount of lean body mass as measured by whole-body DXA scan.
Sustainability of effects of semaglutide on quantity of total right psoas muscle | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the amount of total right psoas muscle as measured in area via CT scan.
Sustainability of effects of semaglutide on quality of abdominal fat (total, subcutaneous, visceral) | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the quality of abdominal fat (total, subcutaneous, visceral) as measured by density via CT scan.
Sustainability of effects of semaglutide on quality of pericardial fat | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the quality of pericardial fat as measured by density via chest CT scan.
Sustainability of effects of semaglutide on quality of total right psoas muscle | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on the quality/intermuscular fat content of total right psoas muscle as measured in density via CT scan.
Sustainability of effects of semaglutide on anthropometric measurements (weight, waist circumference, waist-to-hip ratio) | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on anthropometric measurements.
Sustainability of effects of semaglutide on glucose metabolism | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on glucose metabolism by assessing oral glucose tolerance, fasting glucose levels, and HgbA1C.
Sustainability of effects of semaglutide on lipoprotein profiles | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on lipoprotein profiles and oxidized LDL levels.
Sustainability of effects of semaglutide on systemic inflammation | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on soluble markers of inflammation and immune activation markers to assess overall level of systemic inflammation.
Sustainability of effects of semaglutide on systemic immune activation | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on cellular markers of inflammation and immune activation markers to assess overall level of systemic immune activation.
Sustainability of effects of semaglutide on insulin sensitivity/resistance | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on soluble markers of inflammation and immune activation markers by assessing insulin levels, HOMA-IR (calculated based on insulin levels and glucose levels), and timed insulin levels as part of a 4-hour mixed meal tolerance test.
Sustainability of effects of semaglutide on gut hormones | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on gut hormones, GIP and GLP-1 levels, by means of a 4-hour mixed-meal tolerance test.
Sustainability of effects of semaglutide on gut integrity | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on gut integrity and microbial translocation (e.g., I-FABP, zonulin-1, LPS).
Sustainability of effects of semaglutide on resting energy expenditure | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on resting energy expenditure by means of indirect calorimetry.
Sustainability of effects of semaglutide on pulse wave velocity | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on pulse wave velocity, a measure of arterial stiffness, as a surrogate measure of cardiovascular disease risk.
Sustainability of effects of semaglutide on EndoPat | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on EndoPat, a measure of endothelial function, as a surrogate measure of cardiovascular disease risk.
Sustainability of effects of semaglutide on coronary artery calcium (CAC) score | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on coronary artery calcium (CAC) score as measured by chest CT scan.
Sustainability of effects of semaglutide on overall cardiovascular disease (CVD) risk | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on overall cardiovascular disease (CVD) risk.
Sustainability of effects of semaglutide on bone | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on bone markers and total bone mineral content as measured by whole-body DXA scan.
Sustainability of effects of semaglutide on dietary intake | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on dietary intake via comprehensive dietary intake assessments.
Sustainability of effects of semaglutide on physical activity | 56 weeks
  Sustainability of effects of semaglutide after treatment discontinuation will be investigated, including a comparison of changes over time between participants who received semaglutide vs. placebo, on physical activity status via comprehensive physical activity assessments.

OTHER OUTCOMES:
Effects of semaglutide on adipokines and natriuretic peptides | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on adipokines and natriuretic peptides to help elucidate the potential mechanism by which GLP-1 may affect metabolic endpoints.
Exploratory investigation of mechanisms of semaglutide effects on outcome measures | 32 weeks
  Outcome measures will be evaluated for possible mechanisms/pathways that help elucidate causal effects of semaglutide in people with HIV/HIV-associated lipohypertrophy.
Effects of semaglutide on neurocognitive scores | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on neurocognitive scores assessed using Cognivue test.
Effects of semaglutide on skin AGE measurements | 32 weeks
  Effects of semaglutide will be investigated, including a comparison of changes over time between participants receiving semaglutide vs. placebo, on skin AGE measurements via AGE Reader instrument.
Sustainability of effects of semaglutide on natriuretic peptides | 56 weeks
  A comparison of changes over time will be made between participants receiving semaglutide vs. placebo in adipokines and natriuretic peptides to help elucidate the potential mechanism by which GLP-1 may affect metabolic endpoints.
Sustainability of effects of semaglutide on neurocognitive scores | 56 weeks
  A comparison of changes over time will be made between participants receiving semaglutide vs. placebo in neurocognitive scores assessed using Cognivue test.
Sustainability of effects of semaglutide on skin AGE measurements | 56 weeks
  A comparison of changes over time will be made between participants receiving semaglutide vs. placebo in skin AGE measurements via AGE Reader instrument.
Investigation of mechanisms of semaglutide effects and sustainability of effects on outcome measures | 56 weeks
  Outcome measures will be evaluated for possible mechanisms/pathways that help elucidate causal effects of semaglutide in people with HIV.
Changes over time in HIV-associated lipohypertrophy | 56 weeks
  All outcome measures will be assessed for changes over time among participants receiving placebo to help determine the natural course of lipohypertrophy in HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Grace A McComsey, MD, Principal Investigator — Case Western Reserve University; Allison R Eckard, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this project is an essential part of our proposed activities and will be carried out to comply with the NIH policy on Sharing Research Data. We wish to make our results available both to the community of scientists interested in HIV infection, immune activation and co-morbidities, as well as to people living with HIV infection. The data generated in this project will be presented at local, national and international conferences and published in peer-reviewed journals in a timely fashion. All final peer-reviewed manuscripts that arise from this project will be submitted to PubMed Central. The PI will work to facilitate any request made for data produced under this proposal upon publication of data, using standard, university-approved material/data transfer agreements.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: after publication
Access Criteria: individual requests will be reviewed by study PIs.

REFERENCES:
- [Derived] Atieh O, Daher J, Abboud M, Wu Q, Sattar A, Baissary J, Koberssy Z, Labbato D, Eckard AR, McComsey GA. Effects of Semaglutide on Cognitive Function in People with HIV: A Randomized Controlled Trial. Clin Infect Dis. 2025 Oct 16:ciaf577. doi: 10.1093/cid/ciaf577. Online ahead of print. PMID 41098140
- [Derived] Funderburg NT, Ross Eckard A, Wu Q, Sattar A, Ailstock K, Cummings M, Labbato D, McComsey GA. The Effects of Semaglutide on Inflammation and Immune Activation in HIV-associated Lipohypertrophy. Open Forum Infect Dis. 2025 Mar 20;12(4):ofaf152. doi: 10.1093/ofid/ofaf152. eCollection 2025 Apr. PMID 40160348
- [Derived] Eckard AR, Wu Q, Sattar A, Ansari-Gilani K, Labbato D, Foster T, Fletcher AA, Adekunle RO, McComsey GA. Once-weekly semaglutide in people with HIV-associated lipohypertrophy: a randomised, double-blind, placebo-controlled phase 2b single-centre clinical trial. Lancet Diabetes Endocrinol. 2024 Aug;12(8):523-534. doi: 10.1016/S2213-8587(24)00150-5. Epub 2024 Jul 1. PMID 38964353